CLINICAL TRIAL: NCT06289868
Title: Evaluation of the Access Anti-HAV and Access Anti-HAV IgM Assays As an Aid in the Diagnosis of HAV Infection, and for Detection of Anti-HAV After Vaccination: EU Clinical Trial Protocol
Brief Title: Access Anti-HAV and Access Anti-HAV IgM Assays EU Clinical Trial Protocol (HAV-EU-11-23)
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-TR23-0222; HAV-EU-11-23 (Other: Beckman Coulter, Inc)
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: HAV
Keywords: Hepatitis A Virus (HAV); IgM antibody to Hepatitis A Virus (HAV IgM); antibody to Hepatitis A Virus
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- At-risk and/or signs and symptoms patients of HAV infection and/or HAV test ordered patients: Frozen leftover serum samples from adult and pediatric patients:
  * From subjects exhibiting either jaundice or elevated total bilirubin or elevated serum ALT enzymes and one or more primary signs and symptoms of hepatitis infection, and/or
  * From subjects at-risk of HAV infection, and/or
  * From subjects for whom laboratory testing for hepatitis A was ordered by their healthcare providers.
  Interventions: Diagnostic Test: Access anti-HAV and Access anti-HAV IgM on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays
- Known anti-HAV IgM positive patients: Frozen serum or EDTA retrospective known anti-HAV IgM positive leftover samples procured from sample vendors .
  These samples are known Positive for HAV IgM AND at least one of the following :
  * Positive HAV PCR result (within the last 28 days) OR
  * Jaundice (clinical assessment OR Total bilirubin result >3.0 mg/dL) OR
  * Elevated ALT result (> 200 IU/L)
  Interventions: Diagnostic Test: Access anti-HAV and Access anti-HAV IgM on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays
- HAV Pre- and post-vaccinated patients: Frozen serum leftovers. A first sample was collected, and the US licensed and CE-marked vaccination series administered. A second sample was collected four (4) to ten (10) weeks after the complete vaccination series has been administered according to vaccine dosing instructions.
  Interventions: Diagnostic Test: Access anti-HAV on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays

INTERVENTIONS:
Diagnostic Test: Access anti-HAV and Access anti-HAV IgM on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays — Samples will be tested by comparing Access anti-HAV assay results to final anti-HAV sample status, and Access anti-HAV IgM results to final anti-HAV IgM status, according to respective instructions for use (IFU) or study guide, as applicable, to determine to determine non-reactive (NR), reactive (R), Negative, Positive or Equivocal (EQ).
  For evaluation of the clinical performance of Access anti-HAV assay, all clinical samples will be tested with the reference assays DiaSorin - LIAISON® Anti-HAV and SIEMENS Healthineers Atellica® IM Hepatitis A Total (aHAVT).
  For evaluation of the clinical performance of Access anti-HAV IgM assay, all clinical samples, except pre- and post-vaccinated patient samples, will be tested with the reference assays Abbott - ARCHITECT® HAVAb-IgM, DiaSorin - LIAISON® Anti-HAV IgM, and SIEMENS Healthineers Atellica IM® Hepatitis A IgM (aHAVM).
  Groups: At-risk and/or signs and symptoms patients of HAV infection and/or HAV test ordered patients; Known anti-HAV IgM positive patients
Diagnostic Test: Access anti-HAV on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays — All samples will be tested pre- and post-vaccination by comparing Access anti-HAV assay results to final anti-HAV status, according to respective instructions for use (IFU) or study guide, as applicable, to determine non-reactive (NR), initial reactivity, and repeat reactivity.
  For evaluation of the clinical performance of Access anti-HAV assay, all clinical samples will be tested with the reference assays DiaSorin - LIAISON® Anti-HAV and SIEMENS Healthineers Atellica® IM Hepatitis A Total (aHAVT).
  Groups: HAV Pre- and post-vaccinated patients

SUMMARY:
The purpose of this study is to evaluate the clinical performance supporting that intended purpose of the Access anti-HAV as an aid in the laboratory diagnosis of HAV infection and for detection of anti-HAV after vaccination and of the Access anti-HAV IgM assay as an aid in the laboratory diagnosis of acute or recent HAV infection, on the DxI 9000 Access Immunoassay Analyzer.

This study will be used to obtain CE mark for both Access anti-HAV and anti- HAV IgM assays.

DETAILED DESCRIPTION:
The objective of this study is to determine the diagnostic accuracy of Access anti-HAV and Access anti-HAV IgM assays on the DxI 9000 Access Immunoassay Analyzer, measured as clinical sensitivity and specificity.

The testing will be performed using banked, de-identified, prospective and retrospective US leftover clinical samples, and fully-anonymized retrospective known anti-HAV IgM positive patient samples procured from sample vendors.

ELIGIBILITY:
Inclusion Criteria:

Subject inclusion criteria for the signs and symptoms (S/S), at risk (A/R), HAV test ordered, and Acute HAV Infection cohorts:

* Subjects ≥ 2 years of age
* Subject or legal guardian has signed the Informed Consent Form (ICF) (a minor may need to sign an Assent Form (AF) if required by IRB)
* Subjects who are willing to donate the required amount of blood
* Subjects qualified for one (1) or more of the following four (4) Cohorts:

  * Signs and symptoms (S/S);
  * At risk (A/R);
  * Presumed S/S or A/R (HAV test ordered) and
  * Acute HAV Infection (known anti-HAV IgM positive samples) - these samples are not subject to the individual informed consent and volume criteria.

Subject inclusion criteria for the vaccination cohort

* Subjects 2 years of age or older
* Subjects able to understand and willing to sign the ICF at both pre and post vaccination time points. Subject or legal guardian has signed the Informed Consent Form (a minor may need to sign an assent form if required by IRB)
* Subjects who are willing to donate the required amount of blood: 30 mL
* Subjects with no signs or symptoms of hepatitis as determined by a medical provider, no history of known exposure to HAV
* Subjects previously unvaccinated for HAV

Exclusion Criteria:

* Subjects who previously participated in the study
* Subjects who have received experimental or investigational drugs or treatments within four weeks of phlebotomy

Note for vaccination study: Subjects were screened for anti-HAV prior to vaccination, if positive they were excluded from the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population is the hepatitis A infection diagnostic population, and pre- and post-HAV vaccinated patients for Access anti-HAV assay only.
  Population will include approximately 1,030 subjects as follows:
  * ≥ 930 samples from adult and pediatric patients were collected as part of the US HAV trial prospective and retrospective sample enrollment :
    * From subjects exhibiting either jaundice or elevated bilirubin or elevated serum ALT enzymes and one or more primary signs and symptoms of hepatitis infection, and/or
    * From subjects at-risk of HAV infection, and/or
    * From subjects for whom laboratory testing for hepatitis A was ordered by their healthcare providers.
  * ≥ 100 retrospective known anti-HAV IgM positive samples.
  In addition, for the Access anti-HAV assay only, at least 60 subjects from the US vaccination study will be tested pre and post vaccination in this EU HAV assay clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 1409 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Access Anti-HAV diagnostic accuracy measured as sensitivity and specificity | Baseline
  The endpoints will be diagnostic accuracy measured as clinical sensitivity and specificity of Access anti-HAV assay compared to final anti-HAV status
Access Anti-HAV IgM diagnostic accuracy measured as sensitivity and specificity | Baseline
  The endpoints will be diagnostic accuracy measured as clinical sensitivity and specificity of Access anti-HAV IgM assay compared to final anti-HAV IgM status.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Cerba Xpert, Frépillon
  - Eurofins Biomnis, Ivry-sur-Seine

IPD SHARING:
Plan to Share IPD: No